CLINICAL TRIAL: NCT01275950
Title: An Intervention Study To Evaluate The Impact Of Direct and Surrogate Advertising And Compliance With The Bill With The Respect To Sale Of Tobacco Products Around Educational Institutes
Brief Title: A Study to Evaluate the Impact of Direct and Surrogate Advertising and Compliance With the Bill With the Respect to Sale of Tobacco Products Around Educational Institutes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Sharmila Pimple, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 647
Record Dates: First submitted 2010-06-11; First posted 2011-01-13 (Estimated); Last update posted 2011-01-13 (Estimated); Status verified 2010-06

CONDITIONS: Assessing and Creating Awareness About the Tobacco Law
Keywords: Tobacco vendor; students; knowledge; attitude; practice; direct advertisements; surrogate advertisements
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Health Education — 1. Implementing the intervention programme designed for creating awareness about harmful effect of tobacco (smoked and smokeless forms) and the current regulation to the shop-owners.
  2. Administering the questionnaire to objectively asses the impact of direct/ surrogate tobacco advertisements influencing student behavior and perception about tobacco and tobacco products.
  3. Implementing the intervention programme designed for creating awareness about harmful effect of tobacco (smoked and smokeless forms) and the current regulation to the students through interactive sessions with students in their respective educational institute.

SUMMARY:
The Project aims at enlisting the outlets selling tobacco in any form and enlisting the tobacco based advertisements (Direct and Surrogate) directed towards the community, within 100 yards of the selected educational institutes and studying their impact on the students of that institute. This will further be followed by an intervention program directed at the outlet owners which entails creating awareness about the harmful effects of tobacco and the existing bill and thereby assessing any change in Knowledge, Attitude and Practice. The results thus obtained will facilitate implementation of the existing Bill.

DETAILED DESCRIPTION:
I. Preparatory Phase

1. Selection of Four Educational Institutions for Intervention by Randomized Stratified Sampling Method.

   Mumbai is divided into four zones as being South Mumbai, North Mumbai, East Mumbai and West Mumbai. We shall enumerate all the institutions in these areas and by randomized stratified sampling we shall select one institution from every area resulting in selection of four educational institutions.
2. Recruitment and Training of Staff This involves the recruitment of project personnel and their training. Training would involve the theoretical and practical teaching about health hazards and legal aspects of tobacco use, collecting information by introducing questionnaire, conducting survey, method of area mapping of 100 yards around the educational institution. They would also be trained in identifying establishments selling tobacco based products, identifying direct and indirect tobacco based advertisements.
3. Preparation of Resource Materials and Questionnaire Formats Resource materials to educate the shop owners would be prepared. Questionnaires would be designed to asses the pre and post intervention knowledge of shop owners regarding harmful effects of tobacco and the anti-tobacco bill. A questionnaire to assess the impact of tobacco based advertisements on them would also be designed.
4. Sector wise mapping Mapping of 100 yards of area around the selected education institutions will be conducted by social workers and health care workers.

II. Activity Phase

1. Enlisting of Tobacco/Tobacco Products Selling Establishments within 100 Yards of an Educational Institution
2. Enlisting of Advertisements (direct or indirect) Within 100 yards of an Educational Institution The above two activities will be conducted by social workers and healthcare workers. They would survey 100 yards around the selected institution for area mapping and enlisting the hoardings or any other form of advertisements of tobacco or tobacco based products and shops where these products are sold.

A. Pre-Intervention Phase

1. Observation of compliance with the law. This would involve observation of compliance with the law with respect to presence of signage at the shops as per the current regulations.
2. Awareness Assessment. Assess awareness of shopkeepers (selling tobacco or tobacco based products) about the harmful effects of tobacco and anti-tobacco law regarding sale of tobacco products.

Here a questionnaire would be administered to the shopkeepers to assess their KAP regarding harmful effects of tobacco and tobacco based products and the law.

B. Intervention Phase

1. Implementing the intervention programme designed for creating awareness about harmful effect of tobacco (smoked and smokeless forms) and the current regulation to the shop-owners.
2. Administering the questionnaire to objectively asses the impact of direct/ surrogate tobacco advertisements influencing student behavior and perception about tobacco and tobacco products.
3. Implementing the intervention programme designed for creating awareness about harmful effect of tobacco (smoked and smokeless forms) and the current regulation to the students through interactive sessions with students in their respective educational institute.

C. Post-Intervention Phase

1. Administering the questionnaire to objectively asses the impact of intervention programme on the shop owners of tobacco and tobacco products selling outlets.

III. Evaluation Phase

Outcome measures:

1. The proportion of direct to surrogate advertisements.
2. Compliance of the educational institute with the Tobacco Bill.
3. The proportion of surrogate advertisements which could be recalled with the original tobacco brand, by the students of the selected educational institute.

Pre-assessment and post-assessment of the impact of the intervention programme on the enlisted shop-owners regarding the knowledge, attitude and practices regarding tobacco sale.

ELIGIBILITY:
Inclusion Criteria:

Shop owners of the outlets selling tobacco/ tobacco based products, the outlets lying within 100 yards radius of the selected educational institute.

Students in the age- group of 18-25 years from within the selected educational institute.

Exclusion Criteria:

Students outside the 18-25 yrs age group

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
KAP of tobacco vendors about Tobacco Bill | one year
  The primary outcome is assessment of the Knowledge, Attitude and Practice of shop owners towards tobacco ill-effects and the existing Bill and to determine the impact of our intervention on their knowledge regarding the same. Evaluation of the impact these outlets and the advertisements on the students of the selected educational institutes.

SECONDARY OUTCOMES:
post-intervention KAP | six months
  To evaluate the change in the knowledge attitude and practice six months after our planned intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila A Pimple, MD, Principal Investigator — Tata Memorial Hospital; Gauravi A Mishra, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India